CLINICAL TRIAL: NCT01800734
Title: Absorption and Utilization of a Mixed Meal in Type 1 Diabetes: Creation of a Biological and In Silico Biobank for the Optimization of Artificial Pancreas Systems. A Pilot Study.
Brief Title: Mixed Meal Test in Type 1 Diabetes: Optimization of Artificial Pancreas-Pilot Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Universita di Verona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RBonadonna artificial pancreas
Record Dates: First submitted 2013-02-08; First posted 2013-02-28 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2012-08

CONDITIONS: Diabetes Mellitus Type 1
Keywords: Mixed meal test; Insulin pump; Continuous glucose monitoring; Metabolic control analysis; Closed loop control; Artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clamp-Mixed Meal Arm (Other): Twenty adults patients with type 1 diabetes, regularly attending the Division of Endocrinology and Metabolic Diseases of University of Verona School of Medicine, using continuous subcutaneous fast insulin analogue infusion (CSII) through a permanent pump and on subcutaneous glucose sensing will be enrolled.
  Interventions: Other: Clamp-Mixed Meal Arm

INTERVENTIONS:
Other: Clamp-Mixed Meal Arm — Standard clinical parameters will be assessed in all patients.
  Metabolic tests:
  A. Euglycemic insulin clamp. A standard euglycemic insulin clamp will be carried out to assess insulin sensitivity, as previously described (1).
  B. Mixed meal test. All participants will ingest a standardized mixed meal and will be monitored for 300 minutes thereafter. Right before meal ingestion, a s.c. fast insulin analogue bolus will be administered by the pump
  This test will determine the time courses of:
  1. plasma glucose, 2.13C/12C glucose ratio (hence, meal-derived and endogenous glucose), 3. insulin, 4. free fatty acids, 5. aminoacids, 6. glucagon, 7. incretin hormones 8. glucose control coefficients (CCs) during a mixed meal.

SUMMARY:
Physiology studies will be performed in patients with type 1 diabetes to define during a standardized mixed meal test: 1. The relationship between fast insulin analogue administration by i.v. infusion or by subcutaneous pumps and plasma insulin concentration and tissue insulin action; 2. The relationship between insulin action, glucose fluxes and glucose concentration, the latter one as measured in plasma or estimated by a s.c. glucose-sensor; 3. The concentration curves of some potential modifiers of the glucose-insulin system (i.e.: glucagon, incretin hormones, free fatty and amino acids).

On the basis of these data, in silico phenocopies of the patients (virtual patients) will be created to measure the glucose control coefficients, which quantify the role played by each component of the glucose-insulin system on glucose concentration.

One final purpose of this research is to develop and to optimize an algorithm able to integrate continuous glucose monitoring with continuous subcutaneous fast insulin analogue infusion, known as closed-loop control (CLC) or artificial pancreas.

DETAILED DESCRIPTION:
The maintenance of close-to-normal blood glucose levels slows the onset and progression of long-term microvascular, and possibly macrovascular, complications in patients with type 1 diabetes. Artificial pancreas or integrated CLC [a CLC algorithm which takes into account continuous glucose monitoring (CGM) readings and the effects of previous insulin infusions to continuously compute the amount of insulin dose to be administered] aims to minimize, in real time, glucose variability and prevent extreme glucose excursions (hypoglycemia and hyperglycemia). Despite important developments in sensor and pump technology, the artificial pancreas system must cope with anatomical and functional barriers other than the ones encountered by the normally functioning glucose-insulin system in physiology. For instance , CGM devices measure glucose concentration in the interstitium, not in the blood compartment, introducing a time lag due to glucose diffusion from plasma to the interstitial fluid. Furthermore, insulin (actually, one of current fast insulin analogues) is delivered into the subcutaneous adipose tissue, not in blood, and directly accesses the systemic, not the portal circulation. Owing to these hindrances, developing a smart and suitable CLC algorithm still is an ongoing process. This research aims to alleviate these shortcomings by carrying out clinical physiology study aiming at improving development and optimization of a suitable control algorithm.

Twenty adults patients with type 1 diabetes, regularly attending the Division of Endocrinology and Metabolic Diseases of University of Verona School of Medicine, using continuous subcutaneous fast insulin analogue infusion (CSII) through a permanent pump and on subcutaneous glucose sensing will be enrolled.

Inclusion criteria (see below for more details) are diagnosis of type 1 diabetes as defined by WHO for at least 12 months or confirmed C-peptide negative. Exclusion criteria are recurrent severe hypoglycemia unawareness or clinically significant nephropathy, neuropathy, or proliferative retinopathy.

Standard clinical parameters will be assessed in all patients. Metabolic tests will be carried out at the Division of Endocrinology and Metabolic Diseases of University of Verona School, starting at 08:00 a.m. on two separate days in random order and after a 10-12-h overnight fast. Two metabolic tests will be performed: a euglycemic insulin clamp and a standardized mixed meal test.

A. Euglycemic insulin clamp. A standard euglycemic insulin clamp will be carried out to assess insulin sensitivity, as previously described (1). Subjects will be instructed to use their usual nocturnal fast insulin analogue basal rate, to be left unchanged for at least five hours before the beginning of the test. A CGM device will be inserted two days before the test and calibrated with capillary blood glucose (measured by glucometer) at pre-established hours of the day. Human insulin concentration will be raised with an i.v. prime (0.8 U/m^2 BSA) and maintained constant by an i.v. infusion (40 mU/min·m^2 BSA). Plasma glucose will be allowed to fall until it reaches the physiologic range (i.e. < 5.6 mmol/L), after which it will be clamped at 5.0 mmol/L for at least 60 min by appropriately changing an intravenous infusion of 20% dextrose. Glucose will be measured at bedside by a YSI Glucose Analyzer. Blood samples will be collected at timed intervals to measure plasma insulin (both fast analogue and human insulin), free fatty acids, and glucagon. Continuous glucose (interstitial glucose) monitoring will be performed throughout the insulin clamp.

B. Mixed meal test. This test will be performed to assess the pathophysiology of glucose control during a standardized physiologic challenge. Subjects will be on an Indian corn free and cane sugar free diet for at least one week before study and will be instructed to use the usual nocturnal fast insulin analogue basal rate, to be left unchanged for at least five hours before the beginning of the test. A CGM device will be in place and properly working throughout the test. All participants will ingest a standardized mixed meal (292 Kcal, 38,9 g carbohydrates, 8,9 g fats and 14 g proteins), under the form of maize polenta plus seasoned Italian parmesan cheese, and will be monitored for 300 minutes thereafter. Right before meal ingestion, a s.c. fast insulin analogue bolus will be administered by the pump, according to individual insulin-to-carbohydrate ratio and correction dose. The 13C/12C ratio of maze starch is different from other carbohydrate sources and allows the detection of polenta-derived glucose in the circulation. Plasma glucose, free fatty acid, amino acid, insulin, glucagon, and incretin hormone concentrations will be assessed at baseline and during the entire test. The plasma 13C/12C glucose ratio throughout the test will be monitored by isotope ratio mass spectrometry. CGM data will be collected. This test will determine the time courses of plasma glucose, 13C/12C glucose ratio (hence, meal-derived and endogenous glucose), insulin, free fatty acids, aminoacids, glucagon, and incretin hormones during a mixed meal.

In both studies, blood samples will be put in ice and quickly spun at 1500 g at +4°C. Plasma/serum will be collected and stored at -80°C. Both tests (insulin clamp and mixed meal) will form the biological biobank of this study.

The combined analysis of insulin clamp and mixed meal test data will allow to build a comprehensive model of the glucose insulin system during a mixed meal test in each subject, thereby resulting into an in silico virtual patient, according to a well established methodology developed in our laboratory. The collection of virtual patients with type 1 diabetes undergoing a mixed meal test will form the in silico biobank derived form this study. Virtual patients will be used to carry out Metabolic Control Analysis (MCA), i.e. to compute glucose control coefficients (CCs), which quantify the role played by each component (e.g.: absorption rate of the fast insulin analogue, carbohydrate absorption through the gut, etc.) of the system in determining glucose concentration at each time point during the mixed meal in patients with type 1 diabetes, in close parallelism to the analysis previously carried out by us in patients with type 2 diabetes undergoing an intravenous glucose tolerance test (2). Furthermore, the incretin hormone, glucagon and substrate response to a mixed meal will be quantified, allowing the putative identification of further modifiers of the glucose-insulin system (one for all: glucagon). This database will be instrumental in devising a control algorithm able to guarantee a normal glucose regulation during a mixed meal in patients with type 1 diabetes with CGM on insulin pump therapy.

ELIGIBILITY:
Inclusion Criteria:

* patient must be aged between 18 (inclusive) and 65 years old;
* patient must have been diagnosed with type 1 diabetes(positive islet cell antibodies;
* use of an insulin pump to treat his/her diabetes for at least 1 year;
* actively using a carbohydrate/insulin ratio for insulin bolus adjustments in order to keep blood glucose in a predefined range;
* patient HbA1c is between 6,0% and 9,0% (standardized with DCCT);
* patient must be willing to avoid consumption of acetaminophen containing products during the study involving DexCom (one CGM system which will be employed in this study) use;
* patient must demonstrate proper mental status and cognition for the study;
* patient has signed informed consent from prior to study entry.

Exclusion Criteria:

* diabetic ketoacidosis within the 6 months prior to enrollment;
* severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment;
* pregnancy and breast feeding;
* uncontrolled microvascular (diabetic)complications (other than diabetic non-proliferative retinopathy)such as history of laser coagulation, proliferative diabetic retinopathy, known diabetic nephropathy (other than microalbuminuria with normal creatinine) or neuropathy requiring treatment;
* uncontrolled arterial hypertension (diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg);
* conditions which may increase the risk of hypoglycemia such as uncontrolled coronary artery disease during the previous year (e.g. history of myocardial infarction, acute coronary syndrome, therapeutic coronary intervention, coronary bypass or stenting procedure, stable or unstable angina, episode of chest pain of cardiac etiology with documented EKG changes, or positive stress test or catheterization with coronary blockages >50%), congestive heart failure, history of cerebrovascular event, seizure disorder, syncope, adrenal insufficiency, neurologic disease or atrial fibrillation;
* drugs affecting glucose metabolism (oral steroids, thiazide diuretic, beta-blockers,beta-agonist, nicotinic acid, immunosuppressant agents, antiretroviral drugs and antipsychotics);
* impaired hepatic function measured as alanine aminotransferase or aspartate aminotransferase > three times the upper reference limit;
* impaired renal function measured as creatinine >1.2 times above the upper limit of normal;
* anticoagulant therapy other than aspirin;
* known current or recent alcohol or drug abuse;
* psychiatric disorders that would interfere with study tasks (e.g. inpatient psychiatric treatment within 6 months prior to enrollment);
* mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
1. Composite plasma glucose and hormone responses to a mixed meal 2. Glucose control coefficients | 24 months
  1. Timed curves of composite plasma glucose, meal-derived glucose, endogenous glucose, insulin, glucagon and incretin hormone concentrations in response to a mixed meal
  2. Composite glucose control coefficients (CCs) of each component of the glucose-insulin system at each time point of the mixed meal

SECONDARY OUTCOMES:
Composite plasma free fatty and amino acid responses to a mixed meal | 24 months
  Composite timed curves of plasma free fatty and amino acid concentrations to a mixed meal

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo C Bonadonna, Assoc Prof, Principal Investigator — Division of Endocrinology and Metabolic Diseases, University Hospital of Verona; Enzo Bonora, Full Prof, Study Director — Division of Endocrinology and Metabolic Diseases, University Hospital of Verona; Maddalena Trombetta, Asst Prof, Study Chair — Division of Endocrinology and Metabolic Diseases, University Hospital of Verona
Locations (1):
- Division of Endocrinology and Metabolic Diseases - University Hospital of Verona-Piazzale Stefani 1, Verona, Italy

REFERENCES:
- [Background] Bonetti S, Trombetta M, Boselli ML, Turrini F, Malerba G, Trabetti E, Pignatti PF, Bonora E, Bonadonna RC. Variants of GCKR affect both beta-cell and kidney function in patients with newly diagnosed type 2 diabetes: the Verona newly diagnosed type 2 diabetes study 2. Diabetes Care. 2011 May;34(5):1205-10. doi: 10.2337/dc10-2218. Epub 2011 Mar 16. PMID 21411509
- [Background] Trombetta M, Boselli L, Cretti A, Cali A, Vettore M, Caruso B, Dorizzi R, Avogaro A, Muggeo M, Bonora E, Bonadonna RC. Type 2 diabetes mellitus: a disease of the governance of the glucose-insulin system: an experimental metabolic control analysis study. Nutr Metab Cardiovasc Dis. 2013 Jan;23(1):23-30. doi: 10.1016/j.numecd.2011.05.006. Epub 2011 Sep 19. PMID 21937205